CLINICAL TRIAL: NCT01830491
Title: Comparison of Antiplatelet Effect and Safety of Clopidogrel Napadisilate With Clopidogrel Bisulfate in Coronary Artery Disease Patients: Multi-center, Randomized, Double-blind, Phase IV Clinical Trial
Brief Title: Comparison of Effect & Safety of Clopidogrel Napadisilate With Clopidogrel Bisulfate in Coronary Artery Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-CPG-401
Record Dates: First submitted 2013-04-05; First posted 2013-04-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel napadisilate (Experimental): aspirin 100mg
  Interventions: Drug: Clopidogrel; Drug: aspirin 100mg
- clopidogrel bisulfate (Active Comparator): aspirin 100mg
  Interventions: Drug: Clopidogrel; Drug: aspirin 100mg

INTERVENTIONS:
Drug: Clopidogrel
  Other Names: Pidogul®; Plavix®
Drug: aspirin 100mg

SUMMARY:
The aim of this study is to demonstrate that the combination therapy of aspirin and clopidogrel napadisilate is not inferior to that of aspirin and clopidogrel bisulfate with respect to its effectiveness in inhibiting platelet aggregation, if it is given for four weeks to Coronary Artery Disease (CAD) patients who had been treated with a drug-eluting stent before > 12 months and had remained in a stable condition with a single antiplatelet agent, aspirin.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 to 80 years
* men and women with coronary artery disease who had been treated with drug-eluting stent placement before > 12 months
* patients who had remained in a stable condition with a single antiplatelet agent, aspirin
* patients who did not show any sign or symptom of the worsening of their angina within the last six months that required a coronary artery intervention, a coronary artery bypass, or coronary angiography

Exclusion Criteria:

* Patients who were taking another antiplatelet or anticoagulant drug such as clopidogrel, warfarin, or cilostazol in addition to aspirin, unless they could withdraw from such other drug/s, in which case they could be enrolled in the study after a two-week wash-out period
* Patients who were suffering from drug abuse or alcohol addiction
* hypersensitivity to clopidogrel or aspirin
* severe liver disease (ALT or AST ≥ 10 times the upper normal limit)
* active hemorrhage such as gastro-intestinal ulcer or intracranial hemorrhage
* a high risk of bleeding (blood coagulation disorder, uncontrolled severe hypertension, active bleeding, or history of severe bleeding)
* pregnant or lactating women
* women with childbearing potential who were not using an appropriate contraception method
* had medical or mental contra-indications to the study treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
the percent inhibition of the platelet aggregation change | baseline and 4weeks

SECONDARY OUTCOMES:
the change of P2Y12 reaction unit (PRU) | baseline and 4weeks

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, MD, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Lee HY, Park KW, Kang HJ, Koo BK, Kim HS, Choi DJ, Kim MA, Oh BH. Comparison of antiplatelet effect and safety of clopidogrel napadisilate with clopidogrel bisulfate in coronary artery disease patients: multi-center, randomized, double-blind, phase IV, non-inferiority clinical trial. Am J Cardiovasc Drugs. 2013 Dec;13(6):413-24. doi: 10.1007/s40256-013-0039-y. PMID 23913405